CLINICAL TRIAL: NCT00695344
Title: Prospective and Randomized Study to Evaluate the Effect of Everolimus in the Clinical and Intra-Cardiac Ecography Progression of Heart Graft Vascular Illness.
Brief Title: Study to Evaluate Effect of Everolimus in Progression of Graft Vascular Illness on Patients With Heart Transplant
Acronym: EVEROSTAT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fundacion Investigacion y Desarrollo (Other)
Responsible Party: Dr. Javier Segovia, Hospital Puerta de Hierro
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EVEROSTAT
Record Dates: First submitted 2008-06-09; First posted 2008-06-11 (Estimated); Last update posted 2009-01-30 (Estimated); Status verified 2009-01

CONDITIONS: Cardiac Transplant
Keywords: Effect of everolimus in graft vascular cardiac illness
MeSH Terms: interventions — Everolimus; Azathioprine; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Everolimus 2 times per day + cyclosporin low dose +/- steroids
  Interventions: Drug: everolimus
- 2 (Active Comparator): Cyclosporin + azathioprine or mofetil mycophenolate +/- steroids (the same treatment that patient had before the study).
  Interventions: Drug: azathioprine or mycophenolate mofetil

INTERVENTIONS:
Drug: everolimus — Everolimus 2 times per day, v.o., 2 years treatment.
  Other Names: Certican
  Arms: 1
Drug: azathioprine or mycophenolate mofetil — 2 times per day during 2 years
  Other Names: Imurel; Cellcept
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate if there is a significantly less incidence of major clinical events due to graft vascular illness in recipients of a cardiac transplant on treatment with an immunosuppressive combination, which includes Everolimus, compared to those that continue the previously used immunosuppressive treatment.

DETAILED DESCRIPTION:
This is a prospective, randomized, multicentre, open and controlled study, to evaluate the efficacy and safety of everolimus combined with cyclosporin for microemulsion and steroids according to medical judgement, opposite to the usual therapy which the patient already has received (typically: ciclosporin + azathioprine or mycophenolate mofetil + steroids according to the judgement of the doctor) for patients receiving a cardiac orthotopic transplant since at least 12 months. The patients will be randomized in a 2:1 proportion (everolimus:control), in order to make it possible for the majority of patients to receive the potentially active treatment in a lethal illness for which there is not efficient known treatment up to date.

The study duration will be 2 years of follow-up for each patient. At the end of this period, the patients will be offered the possibility to maintain the immunosuppressive treatment to which they have been assigned, and periodic revisions will be made each 3-6 months.

The two treatment groups are:

Group I - Everolimus twice a day v.o. + cyclosporin for microemulsion in reduced doses +/- steroids.

Group II - Cyclosporin for microemulsion + azathioprine or mycophenolate mofetil +/- steroids (the same administration schedule and medication which the patient received earlier).

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering a heart transplantation at least 12 months before the inclusion.
* Patients with significant graft vascular cardiac illness.

Exclusion Criteria:

* Patients who received more than one solid organ.
* Hypersensibility to everolimus.
* Patients with expected surviving less than 6 months.
* Analytic abnormality significant (platelets < 70.000 plat./mm3, WBC<4.000./mm3, creatinine > 2,5 mg/dl)
* Neoplasm and/or severe systemic illness.
* Mental significant illness.
* Patients who have received sirolimus or everolimus in any moment after transplant.
* Pregnant or lactating woman.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2006-01; Primary Completion 2010-06 (Estimated); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
Percentage of subjects that present at least one major clinical event due to graft vascular illness during the first year of the study on both treatment arms. | December 2010

SECONDARY OUTCOMES:
Intra-coronary ultrasound, safety and adverse events, Nt-proBNP, left ventricular systolic function, coronary stenosis. | December 2010

CONTACTS AND LOCATIONS:
Overall Officials: Javier Segovia, cardiologist, Principal Investigator — Hospital Puerta de Hierro; Nicolás Manito, Cardiologist, Principal Investigator — Hospital Universitari de Bellvitge; Gregorio Rábago, Cardiologist, Principal Investigator — Clínica Universitaria de Navarra; Francisco González-Vílchez, Cardiologist, Principal Investigator — Hospital Marqués de Valdecilla; Juan Delgado, Cardiologist, Principal Investigator — Hospital 12 de Octubre; Juan Fernández Yañez, Cardiologist, Principal Investigator — Gregorio Marañón Hospital; Sonia Mirabet, Cardiologist, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau; Eulalia Roig, Cardiologist, Principal Investigator — Hospital Clinic of Barcelona
Locations (8):
- Spain (8):
  - Hospital Clinic de Barcelona, Barcelona, Barcelona
  - Hospital Santa Creu i Sant Pau, Barcelona, Barcelona
  - Hospital de Bellvitge, Barcelona, Barcelona
  - Hospital Marqués de Valdecilla, Santander, Cantabria
  - Hospital Gregorio Marañón, Madrid, Madrid
  - Hospital Puerta de Hierro, Madrid, Madrid
  - Hospital 12 de Octubre, Madrid, Madrid
  - Clínica Universitaria de Navarra, Pamplona, Navarre